CLINICAL TRIAL: NCT06810219
Title: Cognixion ALS BCI Longitudinal Study
Brief Title: Augmented Reality BCI Longitudinal Study for Persons With Late Stage ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cognixion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ALSUS1
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: usability study; augmented reality; brain computer interface; Amyotrophic lateral sclerosis; als; generative AI; longitudinal study
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Usability Study (Experimental): Participants will utilize the Cognixion Axon-R device and associated communication software for practice and communication tasks as prescribed by the study administrator.
  Interventions: Device: Cognixion ONE

INTERVENTIONS:
Device: Cognixion ONE — A wearable augmented reality brain computer interface with self contained computer and software to enable communication using the device input and output capabilities.

SUMMARY:
The goal of this study is refine the usability of a BCI based communication platform.

The study will take place in the greater Los Angeles area and will enroll up to 10 participants with late stage ALS. Each subject will receive a Cognixion Axon-R augmented reality brain computer interface and associated communication software. The study duration is 3 months for each participant.

The key questions that will be addressed in this study are:

1. How quickly can participants learn and gain confidence with a pure BCI interface.
2. How effective are alternate input modalities including eye tracking for this use case.
3. Identify the extent to which generative AI based personalization impacts the communication quality.

Key measures include:

ITR - information transfer rate SUS - system usability scale

ELIGIBILITY:
Inclusion criteria:

* Must have someone (LAR) who can consent to their participation and who will be present in the study alongside the participant
* Must have a designated individual who can be trained on the Cognixion system
* Fluent in understanding English
* 18 years or older
* Must have ALS and need an assistive communication device
* Must be able to engage in volitional eye opening and sustain eye opening independently for x duration
* Must have a way to communicate apart from using the Cognixion device such as vocalizations, head nod, eye blinks, eyebrow raises, etc. At a minimum, reliable way of communicating "Yes" and "No"

Exclusion criteria:

* Disruption in English comprehension, either due to lack of fluent proficiency or due to a developmental/acquired language disorder (e.g. aphasia)
* Severely hearing impaired or deaf
* Sensitivity to flashing lights
* History of epilepsy and/or seizures
* Vision disorders restricting the visual field such as glaucoma, diplopia (double vision), nystagmus (involuntary eye movements)
* History of vertigo or other vestibular disorders
* Scalp that is prone to irritation, inflammation, injury, or infectious process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
System Usability Score | 3 months from training and setup of device.
  A score ranging from 0 to 100 that captures the usability the device. This is an essential characteristic of a device feasibility study.
Information Transfer Rate (ITR) | 3 months from training and setup of device.
  The rate, in bits per minute, of information transfer for each of the device modalities.
  ITR is measured using a standardized selection procedure.

SECONDARY OUTCOMES:
Words per Minute (WPM) | 3 months from training and setup of device.
  WPM is the number of words that a participant can speak in one minute. This statistic is calculated by counting the total time from partner utterance until a response is spoken by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Principal Investigator, Principal Investigator — Cognixion
Locations (1):
- Cognixion, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Usability insights related to this use case on this type of device will be shared with other accessibility and BCI researchers at conference events and through publications.

REFERENCES:
- [Background] Lewis, J. R. (2018). The System Usability Scale: Past, Present, and Future. International Journal of Human-Computer Interaction, 34(7), 577-590
- [Background] Kellmeyer P, Grosse-Wentrup M, Schulze-Bonhage A, Ziemann U, Ball T. Electrophysiological correlates of neurodegeneration in motor and non-motor brain regions in amyotrophic lateral sclerosis-implications for brain-computer interfacing. J Neural Eng. 2018 Aug;15(4):041003. doi: 10.1088/1741-2552/aabfa5. Epub 2018 Apr 20. PMID 29676287
- [Background] Wolpaw JR, Bedlack RS, Reda DJ, Ringer RJ, Banks PG, Vaughan TM, Heckman SM, McCane LM, Carmack CS, Winden S, McFarland DJ, Sellers EW, Shi H, Paine T, Higgins DS, Lo AC, Patwa HS, Hill KJ, Huang GD, Ruff RL. Independent home use of a brain-computer interface by people with amyotrophic lateral sclerosis. Neurology. 2018 Jul 17;91(3):e258-e267. doi: 10.1212/WNL.0000000000005812. Epub 2018 Jun 27. PMID 29950436